CLINICAL TRIAL: NCT04655144
Title: Intra-Arterial Dexamethasone for the Alleviation of Pain and Postembolization Syndrome Following Uterine Artery Embolization
Brief Title: Dexamethasone for Post Uterine Artery Embolization Pain
Acronym: Dex-Fib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Prasoon Mohan, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200788
Record Dates: First submitted 2020-12-02; First posted 2020-12-07 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: Leiomyoma
Keywords: Fibroids; Leiomyoma; post-embolization pain; dexamethasone
MeSH Terms: conditions — Leiomyoma | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone Arm (Experimental): A total of 5mg dexamethasone will be administered into each uterine artery (10mg total) prior to uterine artery embolization.
  Interventions: Drug: Dexamethasone
- Saline Arm (Placebo Comparator): A volume of normal saline, equal to the total volume delivered in the Dexamethasone Arm, will be administered into each uterine artery prior to uterine artery embolization.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone delivered to the uterine arterial bed, prior to embolization.
  Arms: Dexamethasone Arm
Drug: Saline — Saline delivered to the uterine arterial bed, prior to embolization.
  Arms: Saline Arm

SUMMARY:
The purpose of this research is to investigate if administration steroids (anti-inflammatory medication) via the uterine arteries during uterine fibroid embolization (A non surgical procedure for treating uterine fibroids by blocking their blood supply) can help reduce the pain, nausea, vomiting, and general feeling of weakness following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Women who meet criteria to undergo uterine fibroid embolization for symptomatic fibroids.

Exclusion Criteria:

* Currently pregnant or actively attempting to conceive
* Those deemed mentally impaired to make their own medical decisions
* Previous documented allergy to dexamethasone
* Those currently taking daily steroids for any reason
* Those with diabetes or deemed to be pre-diabetic
* Those with contraindications for angiography
* Prisoners

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prasoon Mohan, MD, Principal Investigator — University of Miami
Locations (1):
- Sylvester Comprehensive Cancer Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone Arm | Saline Arm
Started | 21 | 21
Completed | 20 | 20
Not Completed | 1 | 1
Not completed — Consumed THC | 1 | 0
Not completed — Unilateral embolization | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Arm | Saline Arm | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores Using the VAS Questionnaire
Description: Pain is measured using a modified Visual Analogue Score (VAS), which has a total score ranging from 0 (no pain at all) to 10 (worst pain).
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexamethasone Arm | Saline Arm
Number analyzed (Participants) | 20 | 20
score on a scale
  Preprocedural | 0.8 (1.5) | 1.3 (2.1)
  Immediate | 4 (3.2) | 6.1 (3.1)
  1 Hour | 6 (3.3) | 6.3 (3.2)
  2 Hours | 5.45 (2.9) | 5.8 (3.1)
  3 Hours | 5 (2.8) | 4.9 (3.2)
  6 Hours | 4.6 (2.5) | 5.9 (3.2)
  9 Hours | 4.4 (3.0) | 5.9 (2.9)
  12 Hours | 4.3 (3.3) | 4.5 (3.2)
  24 Hours | 2.5 (2.4) | 4.2 (2.9)
  48 Hours | 2.7 (3.2) | 5.1 (3.0)
  72 Hours | 3.42 (2.9) | 4.7 (3.0)
  96 Hours | 2.35 (2.4) | 4.5 (3.2)
  168 Hours | 1.7 (2.6) | 2.9 (2.4)

2. Secondary Outcome: Severity of Post-embolization Syndrome Symptoms
Description: Post-Embolization Syndrome (PES) was evaluated using a dedicated PES survey.
  For nausea and vomiting, severity will be scored as follows:
  0 - None
  1. - Mild nausea
  2. - Severe nausea requiring antiemetic medication
  3. - Vomiting A score of 0 represents no symptoms (least severe), while a score of 3 represents the most severe symptoms. The scoring range is 0 to 3.
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexamethasone Arm | Saline Arm
Number analyzed (Participants) | 20 | 20
score on a scale
  Preprocedural | 0 (0) | 0 (0)
  Immediate Postprocedural | 0.1 (0.3) | 0.2 (0.5)
  1 Hour | 0.3 (0.8) | 0.4 (0.7)
  2 Hour | 0.4 (0.8) | 0.5 (0.8)
  3 Hour | 0.4 (0.8) | 0.6 (1.0)
  6 Hour | 0.7 (1.0) | 1.1 (1.2)
  9 Hour | 0.8 (1.2) | 1 (1.2)
  12 Hour | 0.6 (0.9) | 0.4 (0.6)
  24 Hour | 0 (0) | 0.2 (0.5)
  48 Hour | 0.2 (0.4) | 0.4 (0.7)
  72 Hour | 0.3 (0.7) | 0.8 (1.1)
  96 Hour | 0.1 (0.4) | 0.4 (0.7)
  168 Hour | 0.2 (0.5) | 0.1 (0.2)

3. Secondary Outcome: Change in Symptoms
Description: The Fibroid Symptom Score was assessed using the Uterine Fibroid Embolization (UFE) Quality of Life and Symptomatology Survey. This survey evaluates eight symptoms:
  1. Degree of bleeding
  2. Presence of clots
  3. Variation in the duration of periods
  4. Variation in the length of periods
  5. Pelvic pain or pressure
  6. Frequency of daytime urination
  7. Frequency of nighttime urination
  8. Fatigue
  Each symptom is scored from 1 to 5, with higher scores indicating more severe symptoms.
  The table below presents the mean change in score for each symptom after the intervention, compared to the pre-procedure score. Higher positive numbers indicate greater symptom improvement. In this table, the maximum possible change for an individual symptom is +4, and the minimum is -4.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexamethasone Arm | Saline Arm
Number analyzed (Participants) | 20 | 20
score on a scale
  Bleeding | 2.4 (1.5) | 2.3 (1.4)
  Clots | 1.7 (1.3) | 1.8 (0.91)
  Fluctuation | 1.9 (1.2) | 1.9 (1.1)
  Length | 1.6 (1.1) | 1.9 (1.1)
  Pain | 1.8 (1.2) | 2.0 (1.2)
  Polyuria | 2.3 (1.5) | 2.2 (1.5)
  Nocturia | 2.3 (1.6) | 2.1 (1.5)
  Fatigue | 2.5 (1.4) | 1.9 (1.4)

4. Secondary Outcome: Change in Quality of Life
Description: Change in participant quality of life was assessed using the Uterine Fibroid Embolization (UFE) Quality of Life and Symptomatology Survey with a total subsection score ranging from 0-6 with the highest score indicating the worst quality of life from fibroid symptoms and vice versa (6=Terrible and 0=Delighted).
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexamethasone Arm | Saline Arm
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 5.2 (1.4) | 5.5 (1.0)
  3 Month | 2.5 (2.0) | 1.3 (1.8)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dexamethasone Arm | Saline Arm
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/21 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Arm (N=21) | Saline Arm (N=21)
Groin hematoma (Surgical and medical procedures) | 1 (1) | 1 (1) — Small access site groin hematomas at the right common femoral artery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT04655144/Prot_SAP_000.pdf